CLINICAL TRIAL: NCT03514004
Title: Using Information and Communication Technologies to Prevent Suicide Among Secondary School Students in Two Regions of Chile: a Randomized Controlled Trial
Brief Title: Using Information and Communication Technologies to Prevent Suicide in Chile
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Chile (Other)
Collaborators: Ministry of Health, Chile (Other Government)
Responsible Party: Principal Investigator, Rubén Alvarado, Principal Investigator, PhD, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ID16I10060
Record Dates: First submitted 2018-04-08; First posted 2018-05-02 (Actual); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Suicide; Adolescent Behavior
Keywords: Suicide prevention; Information and Communication Technologies; Cluster Randomized Controlled Trial; Latin America
MeSH Terms: conditions — Suicide; Adolescent Behavior; Suicide Prevention

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The ICT-based intervention is known as "Project Clan." Each participant randomized to the intervention group will have access to the web platform and mobile applications of "Project Clan" - a virtual community that seeks to promote adolescent mental health and wellbeing as students interact, express themselves, and resolve concerns, with the support of peers and mental health professionals. During the three-month intervention, participants will have complete anonymity, unless trained psychologists supervising the platform as "community counselors" identify behaviors associated with suicide risk and proceed to follow an established emergency protocol. The counselors will be available to answer community questions and provide support on an individual basis.
  Interventions: Behavioral: ICT-based intervention
- Control (No Intervention): Participants in the control group will also be assigned a username and password to access the website, but they will be met with a user interface that only displays a space to answer the corresponding assessments. In addition to the introductory presentation, they will be given a brochure with information regarding adolescent suicide and wellbeing and tips with regard to seeking help and assisting others. This will include the contact information for a telephone hotline, to ensure they can receive professional help if needed.

INTERVENTIONS:
Behavioral: ICT-based intervention — The ICT-based intervention, known as "Project Clan," includes both a web-platform and a mobile application. Project Clan includes both informational and interactive features, ranging from traditional suicide prevention strategies (e.g., a chat with a psychologist, emergency phone hotline, and tips) that seek to reduce barriers to access quality, useful, and evidence-based information and rapid professional assistance, to components designed to increase interactions between participants and promote a sense of belonging and connection with the other "Clan" members.
  Other Names: Project Clan
  Arms: Intervention

SUMMARY:
A cluster randomized controlled trial (RCT) of a program based on information and communication technologies (ICT) will be conducted to prevent suicide and strengthen mental health among secondary school students in Chile. The program utilizes a web-based platform and a mobile application to cultivate a virtual community to promote mental health protective factors, such as self-esteem and self-expression, and reduce suicide risk. It is based on the principles of peer-support and inclusivity, and it has been inspired by previous studies in Europe and the US. The trial will take place in six public secondary schools in two cities of Chile: Santiago and Rancagua. Schools will be randomly assigned to either intervention or control conditions. Assessment will be conducted at baseline, 3-month (post intervention), and at 5-months (2 month follow-up).

DETAILED DESCRIPTION:
There is increasing concern regarding adolescent suicide in Latin America. Recent mental health policies foster the development and implementation of preventive interventions for suicide. Such initiatives, however, have been scarcely developed, even in countries with solid mental health services, such as Chile. The use of information and communication technologies (ICT) might contribute to create accessible, engaging, and innovative platforms to promote well-being and support for adolescents with mental health needs and suicide risk. Promising evidence from high-income countries has already shown the potential benefits of ICT-based programs but further research is needed, especially in settings with restrained resources. Providing local evidence is crucial for persuading policy makers and other stakeholders, and it will prove crucial in order to widely disseminate and scale up the program, if it is found to be effective.

A cluster randomized controlled trial (RCT) to evaluate an ICT-based program will be conducted to prevent suicide and enhance mental health among adolescents in Chile. Four-hundred high-school students will be recruited from 6 public schools in two regions of Chile. Study procedures will be as follows: 1) design of the intervention model and creation of prototype; 2) selection and randomization of the participating schools; 3) implementation of the 3-month intervention and evaluation at baseline, post-intervention period, and a 2-month follow-up.

The ICT-based program utilizes a web-based platform and a mobile application to cultivate a virtual community to promote mental health protective factors, such as self-esteem and self-expression, and prevent adolescent suicide. To overcome the frequent barriers to help seeking, the program will provide rapid direct access to quality, evidence-based information and real-time assistance from a mental health professional; encourage habits that improve emotional and physical health; facilitate self-monitoring of mental health and personal progress; and promote social integration and participation in community-based activities. The program is based on the principles of peer support and inclusivity, and as such, its name is "Project Clan," in reference to a diverse group of individuals who come together for a common purpose in a welcoming environment. The privacy and anonymity of each "Clan member" will be respected, so that they feel free to openly express themselves and resolve questions about possibly taboo topics related to mental health and suicide. Project Clan includes both informational and interactive features, ranging from traditional suicide prevention strategies (e.g., a chat with a psychologist, emergency phone hotline, and tips) that seek to reduce barriers to access quality, useful, and evidence-based information and rapid professional assistance; to components designed to increase interactions between participants and promote a sense of belonging and connection with the other Clan members.

Suicidal ideation is the primary outcome in this study. Secondary outcomes include negative psychological outcomes (e.g., stigma, depression, anxiety) as well as a number of protective psychological and social factors. Indicators regarding the study implementation process will be also gathered. Pertinent study documents (e.g., research protocol, instruments, informed consent, and informed assent forms) were approved by the Ethics Committee for Human Subjects Research of the Faculty of Medicine, Universidad de Chile.

ELIGIBILITY:
Inclusion Criteria:

- Students who attend participating public high schools in two cities (Santiago and Rancagua) of Chile

Exclusion Criteria:

* Students having visual or physical impairments that are incompatible with the intervention model
* Student having a prior diagnosis of a mental disorder.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 400 (Estimated)
Dates: Start 2018-05-30 (Estimated); Primary Completion 2018-09-30 (Estimated); Study Completion 2018-11-01 (Estimated)

PRIMARY OUTCOMES:
Okasha Suicidality Questionnaire | change from baseline suicidality at 5-month follow up
  Self-administered instrument exploring suicidal ideation and beliefs about suicide. Previously linked to suicide intent, depression, despair, low-self-esteem, impulsivity, and low social support. Item is sensitive to identifying immediate risk for suicide attempt. 4 items (scale 0-3; scale range= 0-12).

SECONDARY OUTCOMES:
Coopersmith Self- Esteem Inventory | change from baseline self-esteem at 5-month follow up
  Self-report scale on self-esteem among youth and adolescents in personal and social contexts. 58 items (scale 0-1).
Barratt Impulsiveness Scale | change from baseline impulsiveness at 5-month follow up
  Self-report scale assessing cognitive, motor, and not planned impulsivity. 30 items (scale 0-4).
General Self-Efficacy Scale | change from baseline self-efficacy at 5-month follow up
  Self-report scale assessing self-efficacy among youth across a number of daily stressors. 10 items (scale 1-3).
Coping Across Situations Questionnaire | change from baseline coping at 5-month follow up
  Self-report scale assessing stress coping strategies among youth. 16 items. (scale 1-5).
Perceived Social Support Scale | change from baseline perceived social support at 5-month follow up
  Self-report scale assessing emotional help and advice among youth. 12 items (scale 1-5)
Social Skills Scale | change from baseline social skills at 5-month follow up
  Self-report scale assessing social skills through self-expression of anger or compliance in different scenarios. 33 items (scale 1-4).
Depression Anxiety Stress scales | change from baseline anxiety-depression-stress at 5-month follow up
  Self-report scale assessing depression, anxiety, and stress symptoms. 21 items (scale 0-3).
Discrimination and Devaluation Scale | change from baseline discrimination-devaluation at 5-month follow up
  Self-report scale assessing awareness of stereotyping attitudes towards mental illness (12 items) (scale 0-3).

IPD SHARING:
Plan to Share IPD: No
Given our commitment to the relevancy of this study, we agree to:
  1. Register this study at ClinicalTrials.gov. This record will be updated at least every 12 months, as required.
  2. Report aggregate results no later than one year after the clinical trial completion date, in a publication.
  Furthermore, the University of Chile (UCH) has an internal policy to ensure that clinical trials comply with University and sponsor policy and regulatory standards.

REFERENCES:
- [Derived] Mascayano F, Schilling S, Tapia E, Santander F, Burrone MS, Yang LH, Alvarado R. Using Information and Communication Technologies to Prevent Suicide Among Secondary School Students in Two Regions of Chile: A Randomized Controlled Trial. Front Psychiatry. 2018 Jun 5;9:236. doi: 10.3389/fpsyt.2018.00236. eCollection 2018. PMID 29922187

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-30): https://cdn.clinicaltrials.gov/large-docs/04/NCT03514004/Prot_SAP_000.pdf